CLINICAL TRIAL: NCT06727188
Title: Clinico Laboratory Study of Unresolving Pneumonia in Children
Brief Title: Atypical Pneumonia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Gamal hussein, Resident pediatric doctor., Assiut University
Other Study IDs: Atypical pneumonia
Record Dates: First submitted 2024-09-07; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Unresolving Pneumonia in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Laboratory as cbc crp — Using laboratory and imaging investigations to help in diagnosis and follow up the cases

SUMMARY:
The goal of this observational study is to learn about causes of unresolved pneumonia in children who take appropriate antimicrobial therapy.

DETAILED DESCRIPTION:
Recurrent pneumonia is defined as two episodes of pneumonia in 1 year or three episodes over any time frame. Non resolving pneumonias are characterized by the persistence of symptoms and roentgenographic abnormalities for more than 1 month. The key step in evaluating the patient referred for recurrent or persistent pneumonia is to review the clinical and radiographic features of the episodes to determine if there is adequate documentation to proceed with treatment. After deciding that a patient has had a persistent episode of pneumonia or the requisite number of recurrent episodes of pneumonia (accompanied by radiographic evidence of pulmonary infiltrates), it is essential to classify the episodes into those involving single or multiple lobes. On the basis of this classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incomplete resolution by 4 weeks despite appropriate antimicrobial therapy.

  * From the age of one month to the age of 6 years old.

Exclusion Criteria:

* *Age of the patient below one month and above 6 years old.

  * Patients with chronic lung diseases.
  * Patients with immunodeficiency.
  * Patient with aspiration pneumonia.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children included in the definition of unresolving pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
studying the prevalence of unresolving pneumonia and determining the underlying ateology . | One year
  Recurrent pneumonia is defined as two episodes of pneumonia in 1 year or three episodes over any time frame. Non resolving pneumonias are characterized by the persistence of symptoms and roentgenographic abnormalities for more than 1 month. The key step in evaluating the patient referred for recurrent or persistent pneumonia is to review the clinical and radiographic features of the episodes to determine if there is adequate documentation to proceed with treatment. After deciding that a patient has had a persistent episode of pneumonia or the requisite number of recurrent episodes of pneumonia (accompanied by radiographic evidence of pulmonary infiltrates), it is essential to classify the episodes into those involving single or multiple lobes. On the basis of this classification.

CONTACTS AND LOCATIONS:
Overall Officials: Maher Mokhtar Ahmed, Professor, Study Director — AssiutUniversity; Ahlam Badawi Ali, Doctor, Study Director — AssiutUniversity
Locations (1):
- Pediatrics hospital AssiutUniversity, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Silva GD, Lamabadusuriya SP, Abeywickrema R. Unresolving pneumonia in a child? Look for an aspirated foreign body. Ceylon Med J. 1996 Dec;41(4):159. No abstract available. PMID 9141762